CLINICAL TRIAL: NCT05925400
Title: Effect of Virtual Reality On IN-Vitro fEcuNdation ouTcomes: a Randomized Controlled Trial (VR-INVENT)
Brief Title: Interest of Virtual Reality in the Management of Anxiety and Pain During Embryo Transfer (ET)
Acronym: VR-INVENT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment rate
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/02
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: IVF; Stress; Anxiety
Keywords: Virtual Reality; Embryo transfer; Pregnancy rate
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ET without RV (No Intervention): Patients who will be randomized to the control group will wait for transfer of a fresh blastocyst on the 5th day of development OR a frozen embryo on the 5th day of development according to the usual service protocol.
- ET with RV (Experimental): The transfer and preparation in the transfer room will be done according to the usual service protocol.
  Exposure to virtual reality environment exposure
  Interventions: Device: Virtual Reality during Embryo Transfer

INTERVENTIONS:
Device: Virtual Reality during Embryo Transfer — Patients randomized to the study group, will be provided with the VR headset. The VR exposure will take place 10-15 minutes before the Embryo Transfer (ET) and a 10 min immersion after the ET
  Arms: ET with RV

SUMMARY:
This study compares the use of virtual Reality versus the usual service protocol for the management of anxiety and pain related to In-Vitro fertilization (IVF) procedure

DETAILED DESCRIPTION:
Medical interventions often cause pain, distress or anxiety for most patients.

The use of music and movies has proven effective in pediatrics.

Virtual Reality (VR) is a newer technology that immerses users in a pleasant, three-dimensional environment via a headset. By distracting patients, this technology can reduce anxiety, discomfort and ultimately pain associated with care.

This randomized monocentric trial compares the effect of the use of VR versus without VR during the transfer of a fresh blastocyst on the 5th day of development OR a frozen embryo on the 5th day of development.

The primary outcome will include clinical pregnancy rate and the secondary outcome focuses on the patient's levels of anxiety and stress.

Data on the level of anxiety and stress will be collected through questionnaires before and after the procedure. Also, clinical pregnancy, defined by the presence of one or more gestational sacs with one or more embryos showing cardiac activity, will be assessed through ultrasons 8 ± 4 weeks after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Will benefit from in vitro Fertilization (IVF or ICSI)
* Aged over 18 and under 43,
* Attempt Rank 1 or 2
* Requiring a transfer of a single fresh blastocyst on the 5th day of development OR a frozen embryo on the 5th day of development
* Having received information and given their consent to participate in accordance with the regulations
* Benefiting from a social security scheme or entitled.

Exclusion Criteria:

* Use of frozen sperm
* Use of testicular sperm
* Fecundation technique used: IMSI
* Early embryo transfer on D2 or D3
* Inability to understand the information given
* Under guardianship, under curatorship or under safeguard of justice,
* Communication difficulties or neuropsychic disorders,
* Current corneal or conjunctival pathologies,
* Claustrophobia,
* Appearance of nausea in the mountains or at sea,
* Regular use of anxiolytics

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | Assessed 12 weeks after embryo transfer
  Clinical Pregnancy Rate defined by the presence of one or more gestational sacs with one or more embryos showing cardiac activity

SECONDARY OUTCOMES:
State and Trait Anxiety Inventory (STAI) questionnaires | Questionnaires will be filled out in 2 different time points during the study: 1) ET day, 45 minutes before ET 2) ET day, 10 minutes after ET procedure
  The rate of anxiety and stress level before and after embryo transfer, measured by the State and Trait Anxiety Inventory (STAI) StAI-Y1-State ranging from 20 to 80 (20 = Low Level of Anxiety), 80 = High Level Of Anxiety) StAI-Y2-Trait ranging from 20 to 80 (20 = Low Level of Anxiety), 80 = High Level Of Anxiety)
Generalized Anxiety Disorder - 7 (GAD-7) questionnaires | Questionnaires will be filled out in 2 different time points during the study: 1) ET day, 45 minutes before ET 2) ET day, 10 minutes after ET procedure
  The rate of anxiety and stress level before and after embryo transfer, measured by Generalized Anxiety Disorder - 7 (GAD-7) questionnaires GAD-7 ranging from 0 to 21 (0= No or Minimal Stress, 21= Worst Possible Stress)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Pierre Cherest, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No